CLINICAL TRIAL: NCT01339221
Title: Epidemiological, Observational, Post Marketing Study of the Genetic Stability of GSK Biologicals' Rotavirus Vaccine (Rotarix™) in Children <5 Years of Age Diagnosed With Severe Gastroenteritis, in Belgium
Brief Title: Epidemiological, Observational and Post Marketing Study of Rotarix™ in Children With Severe Gastroenteritis in Belgium
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112560
Record Dates: First submitted 2011-04-14; First posted 2011-04-20 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Infections, Rotavirus
Keywords: Observational; Rotarix™; post-marketing
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples Without DNA — Stool samples

GROUPS / COHORTS (2):
- Cohort A: Children confirmed with G1 and/or P[8] cases from the RotaBel study
  Interventions: Procedure: Stool samples
- Cohort B: Children hospitalized for severe gastroenteritis in the study hospitals and tested positive for rotavirus
  Interventions: Procedure: Stool samples

INTERVENTIONS:
Procedure: Stool samples — Stool samples collected and checked for the presence of rotavirus

SUMMARY:
The main aim of this study is to investigate cases of rotavirus gastroenteritis in Belgian children with opportunity to receive Rotarix™ to monitor the potential occurrence of genetic drifts (point mutations) in the vaccine strain and the occurrence of genetic shifts (re-assortments) between vaccine and naturally circulating wild-type strains in Belgium population after the introduction of Rotarix™. The study will also detect if there is any alteration in rotavirus pathogenicity conferred by re-assortment and if the mutated vaccine strain is still efficacious in preventing rotavirus gastroenteritis.

DETAILED DESCRIPTION:
This study is conducted in two phases: Phase I and Phase II. Phase I will be retrospective and consist of re-using the data collected in RotaBel (EPI-ROTA-111426) study. Phase II will be prospective and consist of maintaining the active surveillance system to identify rotavirus cases in several hospitals in Belgium.

ELIGIBILITY:
Inclusion Criteria:

Phase I:

• Vaccinated and unvaccinated confirmed G1 and/or P[8] rotavirus gastroenteritis cases from the RotaBel study.

Phase II:

* A male or a female, born after 1 October 2006 and aged between 14 weeks and < 5 years at the time of hospital admission.
* Child admitted at the study hospital for severe gastroenteritis during the study period.
* Onset of severe gastroenteritis ≤14 days prior to admission.
* Child whose stool sample was tested positive for rotavirus by a hospital routine test.
* Written informed consent obtained from the parent or guardian of the child.

Exclusion Criteria:

• Child in care.

Ages: 14 Weeks to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children confirmed with G1 and/or P[8] cases from the RotaBel study, children between 14 weeks and <5 years of age, hospitalized for severe gastroenteritis in the study hospitals and who are tested positive for rotavirus
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of rotavirus gastroenteritis among children hospitalized with acute gastroenteritis who have had opportunity to receive Rotarix™. | Over a three-year period
Occurrence of G1 and/or P[8] rotavirus gastroenteritis among children hospitalized with rotavirus gastroenteritis | Over a three-year period
Occurrence of vaccine-derived G1 and/or P[8] encoding gene segments among children hospitalized with rotavirus gastroenteritis due to G1 and/or P[8] strains | Over a three-year period
Occurrence of mutated vaccine strains and re-assortments among hospitalized children with vaccine-derived G1 and/or P[8] encoding gene segments | Over a three-year period
Clinical characteristics of hospitalized children with vaccine-derived G1 and/or P[8] encoding gene segments, and with vaccine-derived re-assortant strains and vaccine-derived mutated strains | Over a three-year period
  Clinical characteristics include symptoms of current gastroenteritis (GE) episode, severity of GE episode by Vesikari score, date of onset of GE episode, diagnosis at admission, diagnosis at discharge, treatment, medical history and co-infections.
Occurrence of co-infections due to other common viral intestinal pathogens (norovirus, astrovirus, adenovirus) among hospitalized children with rotavirus gastroenteritis | Over a three-year period
Epidemiological characteristics of hospitalized children with vaccine-derived G1 and/or P(8) encoding gene segments, and with vaccine-derived re-assortant strains and vaccine-derived mutated strains | Over a three-year period
  Epidemiological characteristics include age, gender, centre of hospitalization, date of admission, date of discharge, duration of hospitalization, etc.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Belgium (10):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Deurne
  - GSK Investigational Site, Eeklo
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Namur
  - GSK Investigational Site, Roeselaere
  - GSK Investigational Site, Sint-Truiden
  - GSK Investigational Site, Wilrijk